CLINICAL TRIAL: NCT02715375
Title: A Double Blind, Randomized, Sham Controlled Trial to Investigate the Effect of the CREON2000A on Asthma Control in Children With Mild to Moderate Persistent Asthma
Brief Title: Investigate the Effect of the CREON2000A on Asthma Control in Children With Mild to Moderate Persistent Asthma
Acronym: CREON2000A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Innovations and Goods, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Cincinnati (Other); Bernstein Clinical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U44-CRE-01; U44AI074918 (NIH)
Record Dates: First submitted 2016-03-10; First posted 2016-03-22 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Asthma
Keywords: asthma environment
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device: CREON2000A (Experimental): Children with mild to moderate asthma maintains allergy medicines have an experimental ultra violet device installed in their homes.
  Interventions: Device: CREON2000A
- Device: Sham Comparator (Sham Comparator): Children with mild to moderate asthma maintains allergy medicines have a sham device using a shielded blue light sham lamp that otherwise resembles the experimental device installed in their homes.
  Interventions: Device: CREON2000A

INTERVENTIONS:
Device: CREON2000A

SUMMARY:
This is a pivotal, 12-month, randomized, sham controlled, parallel group, multicenter, double blind study with an allocation ratio of 1:1. The study population is children between the ages 6 to 17 years, with mild to moderate persistent asthma. The purpose of the study is to determine whether the CREON2000A, an environmental control device, will decrease asthma severity, as measured by the Composite Asthma Severity Index (CASI), in children with mild to moderate persistent allergic asthma over a twelve month period.

DETAILED DESCRIPTION:
The pilot study (Protocol #PA-01-052; Health Effects of CREON2000 in Asthmatic Children. IB ID# GI 1001) offered preliminary evidence that the CREON2000A system may be beneficial in asthma. This study is a follow-up, using children, aged 6 to 17 with mild to moderate persistent asthma, as the subjects of the study. Children are usually treated with fewer controller medications and have fewer confounding co-morbidities making it more likely to detect a therapeutic benefit from an environmental intervention. The study will involve 4 study site visits, 2 home visits, and 7 phone calls. Adjustment of asthma therapy by the site clinician will occur at baseline (Visit 1) and at each follow-up office visit after Visit 1 using a modified algorithm based on the National Asthma Education and Prevention Program Expert Panel Report 3 (NAEPP EPR3) guidelines. Enrollment will be over 18 months. The study duration for each subject will be 12 months.

ELIGIBILITY:
Inclusion criteria

1. Males and Females ages 6.0 to 17.0 years.
2. Subjects with a physician diagnosis of mild or moderate persistent asthma.
3. FEV1 ≥ 60% predicted with ≥ 12% improvement after bronchodilator therapy.
4. Must have evidence of; 1) serum specific IgE (immunocap) ≥ .35 or 2) a positive skin prick test to one or more common indoor allergens including standardized house dust mite, cat, dog, cockroach, mouse in the past.

Exclusion criteria

1. Current smokers
2. Passive exposure to environmental tobacco smoke at home or active fireplaces and other sources of air particulates (wood burning stoves, kerosene heaters) at home.
3. Diagnosed by a physician with a chronic lung disease other than asthma.
4. Upper or lower respiratory infection within four weeks prior to enrollment.
5. Known to have any other chronic illness (besides asthma) that is not well controlled at the time of screening (Visit 1).
6. History of a life threatening asthma attack requiring cardiopulmonary support, intubation with ventilatory support, hospitalization in an intensive care unit or hospitalization for asthma within 6 months preceding study screening (Visit 1).
7. Participation in another investigational drug/device study within the past 3 months (not including chart or observational studies)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Change in CASI Score | Baseline and 12 months
  Difference between study arms in the change in asthma severity as measured by the Composite Asthma Severity Index (CASI) from Baseline (Visit 1) to the 12-month follow up office visit

SECONDARY OUTCOMES:
Change in Forced Expiratory Volume (FEV1) | Baseline and 12 months
  • in the mean change in FEV1 (% predicted) from Baseline (Visit 1) to 12-month follow up office visit
Mean change in number of day time symptom scores | Baseline, 4, 8 and12 months
  • in the mean change in number of day time symptom scores from Baseline (Visit 1) to the 4, 8 and 12-month follow up office visits
Mean change in number of night time symptoms | Baseline, 4, 8 and 12 months
  • in the mean change in number of night time symptom scores from Baseline (Visit 1) to the 4, 8 and 12-month follow up office visits
Mean change in the number of daily puffs/inhalations of short-acting beta-agonist (SABA) rescue medication | Baseline, 4, 8 and 12 months
  • in the mean change in the number of daily puffs/inhalations of short-acting beta-agonist rescue medication taken over 14 days prior to each evaluation, from Baseline (Visit 1) to 4, 8 and 12 month follow up office visits
Mean Change in CASI | Baseline, 4, 8 and 12 months
  • in the mean change in CASI from Baseline (Visit 1) to 4- and 8- and 12-month follow up office visits
Mean change in daily does of inhaled glucocorticoids taken (µg/day) | Baseline 4, 8 and 12 months
  • in the mean change in daily dose of inhaled glucocorticoids taken (µg/day) by participants from Baseline (Visit 1) to 4, 8 and 12 months follow up office visits.
Mean change in the percentage of patients with an asthma exacerbation | Baseline and12 months
  • in the mean change in the percentage of patients with an asthma exacerbation during the period from baseline (Visit 1) to the 12 month follow up office visit

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bernstein, MD, Study Chair — University of Cincinnati, Cincinnati, Ohio; Mark Glazman, PhD, Principal Investigator — General Innovations and Goods, Inc. (GI&G)
Locations (8):
- United States (8):
  - Advanced Research Institute of Miami, LLC, Homestead, Florida
  - Allergy & Asthma Associates, Lexington, Kentucky
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Columbus Nationwide Children's Hospital, Columbus, Ohio
  - Ohio Pediatric Research Assn., Dayton, Ohio
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Great Lakes Medical Research, LLC, Willoughby, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bernstein JA, Seth A, Rao M, Katz JC, Singh U, Greisner W, Lierl M, Prince B, Mavunda K, Bernstein CK, Guan T, Nation AJ, Rudman Spergel AK, Togias A, Glazman M. Randomized trial of ultraviolet irradiation units installed in homes of children and adolescents with asthma. J Allergy Clin Immunol Glob. 2025 Jan 29;4(2):100427. doi: 10.1016/j.jacig.2025.100427. eCollection 2025 May. PMID 40091880